CLINICAL TRIAL: NCT07123350
Title: Evolving Biologic Administration: Evaluating the Shift From Intravenous to Subcutaneous Vedolizumab for Inflammatory Bowel Disease
Brief Title: Evaluating the Shift From Intravenous to Subcutaneous Vedolizumab for Inflammatory Bowel Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Takeda Pharmaceuticals U.S.A., Inc. (Unknown)
Responsible Party: Principal Investigator, Chelsea Renfro, Clinical Pharmacist for Research and Engagement, Vanderbilt University Medical Center
Other Study IDs: 250579
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn&Amp;#39;s Disease (CD); Ulcerative Colitis (UC)
Keywords: Inflammatory Bowel Disease; Health-system Specialty Pharmacy; Vedolizumab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- IV to SC switch: Patients with Crohn's Disease (CD) or Ulcerative Colitis (UC) referred to switch to subcutaneous vedolizumab from IV vedolizumab from a VUMC IBD provider and receive at least 1 dose of subcutaneous vedolizumab
  Interventions: Drug: Patient switched from IV vedolizumab to subcutaneous vedolizumab as part of normal patient care

INTERVENTIONS:
Drug: Patient switched from IV vedolizumab to subcutaneous vedolizumab as part of normal patient care — This study does not include any subject enrollment or randomization. This is a retrospective cohort review of patients referred to start subcutaneous vedolizumab from a VUMC IBD provider.

SUMMARY:
The goal of this retrospective study is to learn about dosing patterns in patients starting subcutaneous vedolizumab administration and patient outcomes after starting subcutaneous administration.

Patients with IBD who are starting subcutaneous vedolizumab administration between September 1, 2023, and March 31, 2025, as part of normal patient care, will be retrospectively reviewed and analyzed.

DETAILED DESCRIPTION:
Vedolizumab intravenous (IV) infusions have been a first-line treatment option for patients with inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC) for over ten years. Recently, vedolizumab has been approved by the Food and Drug Administration for subcutaneous (SC) administration in the United States, offering patients a more convenient treatment option with medication administration at home. Evidence, largely from European countries where the SC formulation of vedolizumab has been available since 2020, shows a durable and potentially improved clinical response when switching to the SC formulation. A high SC treatment persistence has been found, mainly above 80%. Additionally, many patients accept the transition to SC vedolizumab as a safe and feasible treatment option and noting that the shorter treatment duration was specifically advantageous.

Current evidence is limited by the minimal amount of data on patients transitioning from IV to SC vedolizumab. For treatment with vedolizumab IV to SC, large scale, real-life studies with long term follow-up are necessary. More research is needed to further evaluate predictors for a relapse when transitioning from IV to SC therapy that have been seen in previous studies, including older age, escalated IV dosing, fecal calprotectin >250 microgram/gram at baseline, and CRP > 2g/L at baseline. We must also evaluate patient clinical outcomes after switching from IV to SC vedolizumab or infliximab and potential predictors for a positive response. These results will drive clinical decisions and further understanding of treatment expectations.

There is also a large gap in available information on standard and escalated dosing patterns before and after switching from IV to SC vedolizumab. Minimal research has evaluated whether or not patients on escalated IV dosing maintain escalated dosing at the time of switch or initiate standard SC dosing. There is a pressing need to understand dosing patterns in patients transitioning from escalated IV dosing to SC administration and patient outcomes after switching to SC administration based on dosing.

The proposed study would meet current gaps in literature by evaluating 1) clinical outcomes in patients with CD and UC switching from IV to SC vedolizumab and 2) dosing patterns from standard or escalated IV dosing at baseline to standard or escalated SC dosing, including switching practices and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's Disease or Ulcerative Colitis referred to start SC vedolizumab from a VUMC IBD provider and receive at least 1 dose of subcutaneous vedolizumab
* Age 18 years old or older

Exclusion Criteria:

* Patients prescribed SC vedolizumab from a non-VUMC provider
* Patients lost to follow-up or change in provider or medication before SC formulation started

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were identified if they were seen in the VUMC IBD clinic as part of normal clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission | baseline with IV dosing, and 3, 6, 9, 12 months after switching to SC
  Defined as clinical remission assessed and written by provider in the office visit note

SECONDARY OUTCOMES:
Endoscopic Remission | at baseline with IV dosing and within 12 months after switching to SC
  Endoscopic remission as seen by provider after colonoscopy assessment
Dosing patterns of IV dose/frequency and SC dose/frequency | At baseline and up to 12 months after switching
  standard dosing vs escalated dosing; includes any dose changes of the SC product within 12 months after switching from IV to SC
SIBDQ score | Baseline and 12 months post switch to SC
  Short Inflammatory Bowel Disease Questionnaire: 10-item validated health-related quality of life tool that measures physical, social, and emotional status. It is designed to evaluate how the patient is feeling over the past two weeks. The 10 questions are given scores of 1 to 7 with an overall score of 10 to 70. The lower the score, the more severe the disease is impacting the patient's quality of life (QOL).
Persistence to SC formulation | Up to 12 months after switching
  Measured by time to discontinuation; will include reason for discontinuation if SC stopped
Adverse events to vedolizumab SC | Up to 12 months after switching
  Adverse events to vedolizumab SC that required change back to IV
Adherence | 12 months post switch to SC
  Measured by PDC
Patient-reported missed doses | 12 months post switch to SC
  For patients filling with Vanderbilt Specialty Pharmacy only; will include reasons for patient-reported missed doses
Maintenance steroid use for IBD | 12 months post switch to SC
  Will determine if maintenance steroids were used for maintenance post switch to SC (yes/no)
Number of steroid prescriptions for flares | 12 months before and after switch
  Based on prescription history in patient chart

OTHER OUTCOMES:
Hospitalization and ED visits related to IBD | 12 months before and after switch to SC
  Determined based on visits documented in patient chart
Adverse events reported after switching to SC | 12 months post switch to SC
  Will only be assessed for patients filling with Vanderbilt Specialty Pharmacy
Drug trough levels before and after switching to SC | 12 months before and after switching to SC
  Vedolizumab trough levels

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Z. Kozlicki, PharmD, Principal Investigator — Vanderbilt University Medical Center; Chelsea P. Renfro, PharmD, Principal Investigator — Vanderbilt University Medical Center; Autumn D. Zuckerman, PharmD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Study does not meet the criteria for an Applicable Clinical Trial (ACT) under 42 CFR 11.22(b) as this study is not interventional (a clinical trial)